CLINICAL TRIAL: NCT06411691
Title: Pooled Mutant KRAS-Targeted Long Peptide Vaccine Combined With Balstilimab and Botensilimab for Patients With Stage IV MMR-p Colorectal Cancer and Pancreatic Ductal Adenocarcinoma
Brief Title: KRAS-Targeted Vaccine Combined With Balstilimab and Botensilimab for Patients With Stage IV MMR-p Colorectal Cancer and Pancreatic Ductal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Agenus Inc. (Industry); Private Philanthropic Funds (Other); National Cancer Institute (NCI) (NIH); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J2456; IRB00427416 (Other: Johns Hopkins Medicine IRB); 1R01CA296410-01 (NIH); HT94252410948 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer; Pancreatic Cancer
Keywords: mKRAS peptide vaccines; Anti-PD-1 (anti-check point inhibitor); PD-L1 (check point inhibitor); Balstilimab; Botensilimab; Cancer Vaccines; SLP mKRASvax (peptide vaccine + Poly-ICLC (Hiltonol)); Immunotherapy; Colon Cancer; Metastatic colon cancer; Pancreatic Ductal Adenocarcinoma (PDAC); Metastatic pancreatic cancer; Hiltonol
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms | interventions — poly ICLC; balstilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SLP mKRASvax (Up to 1.8mg peptide + 0.5 mg Poly-ICLC (Hiltonol), Botensilimab and Balstilimab (Experimental)
  Interventions: Drug: KRAS Vaccine with Poly-ICLC adjuvant; Drug: Balstilimab; Drug: Botensilimab

INTERVENTIONS:
Drug: KRAS Vaccine with Poly-ICLC adjuvant — SLP mKRASvax with Poly-ICLC adjuvant will be administered on days 1, 8, 15 and 22 in Cycle 1 (Prime Phase) and on day 1 in cycle 4 and every other cycle and beyond (Boost Phase). Up to 5 subcutaneous injections will be administered in the upper thighs, arms and/or back.
  Drug: 0.3 mg per peptide vaccine + 0.5mg Poly-ICLC
  Other Names: Hiltonol® (Poly-ICLC)
Drug: Balstilimab — 240 mg will be administered as a 30 minute IV. Infusion (-10/+25 minutes) on day 1 and day 15 during Cycle 1 in Prime Phase and on day 1 and day 15 of every cycle in the Boost Phase beginning on Cycle 2 (for a maximum of 2 years from initial vaccination).
  Drug: 240 mg IV
  Other Names: AGEN2034
Drug: Botensilimab — 75 mg will be administered as a 30 minute IV. Infusion (-10/+25 minutes) on Cycle 1 day 1 in Prime Phase and on Cycle 2 day 15 in the Boost Phase.
  Drug: 75 mg IV
  Other Names: AGEN1181

SUMMARY:
Phase 1b study evaluating the efficacy and immune response to a synthetic long peptide mutant KRAS vaccine (SPL mKRASvax) combined with Balstilimab and Botensilimab for unresectable or metastatic mismatch repair-proficient (MMR-p) colorectal cancer (mCRC) or unresectable or metastatic MMR-p pancreatic ductal adenocarcinoma (PDAC) patients with measurable disease following first-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Have histologically or cytologically - proven cancer of the pancreas or colon.
* Have tumor lesions amenable to repeated biopsy, and patient's acceptance to have a tumor biopsy of an accessible lesion at baseline and on treatment if the lesion can be biopsied with acceptable clinical risk (as judged by the investigator).
* Measurable disease as per RECIST 1.1.
* Have sufficient and accessible tissue for next generation sequencing (NGS) and immune-phenotyping.
* Have one of the KRAS mutations included in the vaccine at the time of vaccination expressed in tumor.
* Cohort A: Have received 4-6 months of FOLFIRINOX or gemcitabine+nab-paclitaxel for the 1st line treatment of metastatic unresectable PDAC.
* Cohort B: Have received 4-6 months of 1st line SOC chemotherapy per NCCN guidelines (FOLFIRINOX, FOLFOX, FOLFIRI +/- targeted therapy with VEGFi or EGFRi) of metastatic CRC.
* Cohort C: Have received no more than 3 lines of systemic chemotherapy, including prior KRAS inhibitor.
* Eastern Cooperative Oncology Group (ECOG) performance status 0.
* Life expectancy of greater than 3 months.
* Patients must have adequate organ and marrow function defined by study-specified laboratory tests prior to initial study drug.
* Woman of childbearing potential must have a negative pregnancy test and follow contraceptive guidelines as defined per protocol.
* Men must use acceptable form of birth control while on study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Is a candidate for definitive surgical resection.
* Known history or evidence of brain metastases and/or leptomeningeal spread.
* Prior treatment with immunotherapy agents (including, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA4, etc.).
* Receiving active immunosuppressive agents or chronic use of systemic corticosteroids within 14 days of vaccine treatment.
* Has active autoimmune disease that has required systemic treatment in the past 5 years, or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents.
* Known history or concurrent interstitial lung disease.
* Has a pulse oximetry < 95% on room air.
* Requires the use of home oxygen.
* Infection with HIV or hepatitis B or C.
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, metastatic cancer, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has been diagnosed with another cancer or myeloproliferative disorder in the past 5 years except for superficial bladder cancer, non-melanoma skin cancers, DCIS, a low-grade prostate cancer, or a cancer not expected to impact life expectancy and not requiring therapy.
* Has had surgery within 28 days of dosing of investigational agent, excluding minor procedures (dental work, skin biopsy, etc.), celiac plexus block, and biliary stent placement.
* Has received any non-oncology live vaccine therapy used for prevention of infectious diseases within 28 days of study treatment.
* If at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or other substance abuse (including alcohol) that could potentially interfere with adherence to study procedures or requirements.
* Any other sound medical, psychiatric, and/or social reason as determined by the Investigator.
* Unwilling or unable to follow the study schedule for any reason.
* Are pregnant or breastfeeding.
* Any radiological or clinical pleural effusions or ascites.
* History of malignant small bowel obstruction.
* On parenteral nutrition.
* Known or suspected hypersensitivity to Hiltonol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Cohort A: Progression-free Survival (PFS) for maintenance mPDAC cohort | 4 months
  PFS is defined as the number of mPDAC patients free of progression at 4 months since the initiation of therapy - disease progression (progressive disease [PD] or relapse from complete response [CR] as assessed using RECIST 1.1 criteria) or death due to any cause. Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30percent decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20percent increase in sum of diameters of target lesions, Stable Disease (SD) is <30percent decrease or <20percent increase in sum of diameters of target lesions.
Cohort B: Objective Response Rate (ORR) for maintenance mCRC cohort | 3 years
  ORR is defined as the number of mCRC patients who are administered at least 1 dose of SLP mKRASvax achieving a complete response (CR) or partial response (PR) based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) at any time during the study. CR = disappearance of all target lesions, PR is =>30percent decrease in sum of diameters of target lesions, progressive disease (PD) is >20percent increase in sum of diameters of target lesions, stable disease (SD) is <30percent decrease or <20percent increase in sum of diameters of target lesions.
Cohort C: Objective Response Rate (ORR) for KRAS-inhibitor exposed mPDAC cohort | 3 years
  ORR is defined as the number of mCRC patients who are administered at least 1 dose of SLP mKRASvax achieving a complete response (CR) or partial response (PR) based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) at any time during the study. CR = disappearance of all target lesions, PR is =>30percent decrease in sum of diameters of target lesions, progressive disease (PD) is >20percent increase in sum of diameters of target lesions, stable disease (SD) is <30percent decrease or <20percent increase in sum of diameters of target lesions.
Number of participants experiencing study drug-related toxicities | 3 years
  Number of participants experiencing study drug-related adverse events Grade 3 or higher as defined by CTCAE v5.0

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per RECIST 1.1 | 3 years
  ORR is defined as the number of mPDAC patients who are administered at least 1 dose of SLP mKRASvax and balstilimab +/- botensilimab achieving a complete response (CR) or partial response (PR) based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) at any time during the study. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on the Kaplan-Meier curve.
Disease Control Rate (DCR) | 2 months
  DCR is defined as the number of patients who are administered ≥ 1 dose of SLP mKRASvax achieving a complete response (CR) or partial response (PR) and stable disease (SD) based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) at 2 months post first vaccination. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Disease Control Rate (DCR) | 6 months
  DCR is defined as the number of patients who are administered ≥ 1 dose of SLP mKRASvax achieving a complete response (CR) or partial response (PR) and stable disease (SD) based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) at 6 months post first vaccination. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Disease Control Rate (DCR) | 12 months
  DCR is defined as the number of patients who are administered ≥ 1 dose of SLP mKRASvax achieving a complete response (CR) or partial response (PR) and stable disease (SD) based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) at 12 months post first vaccination. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Progression-free Survival (PFS) per RECIST 1.1 | 3 years
  PFS is defined as the time from cycle 1, day 1 of KRAS vaccine and balstilimab and botensilimab until first documented local disease progression (progressive disease [PD] or relapse from complete response [CR] as assessed using RECIST 1.1 criteria) or death due to any cause. Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Nilofer Azad, MD, Principal Investigator — SKCCC Johns Hopkins Medical Institution
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No